CLINICAL TRIAL: NCT05692804
Title: Evaluation of Intraoperative Neuronal Damage in Patients Undergoing Robot-assisted Laparoscopic Radical Prostatectomy With S100beta, GFAP and NSE Biomarkers
Brief Title: Evaluation of Neuronal Damage in Patients Undergoing Robot-assisted Laparoscopic Radical Prostatectomy With Biomarkers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, İlker Onguc Aycan, PROFFESSOR,MD, Akdeniz University
Other Study IDs: Brain damage in RALRP
Record Dates: First submitted 2023-01-12; First posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Brain Damage; Postoperative; Surgery-Complications
Keywords: brain damage; postoperative; Robot-assisted laparoscopic radical prostatectomy (RALRP); GFAP; NSE; S100B
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group with Sevoflurane: The Sevoflurane used for maintenance of general anesthesia
  Interventions: Diagnostic Test: Mini Mental State Examination(MMSE),Montreal Cognitive Assessment ( MoCA),S100B ( protein S100 subunit beta) ,GFAP ( glial fibrillary acidic protein ),NSE ( neuron-specific enolase )
- Group with Propofol: The Propofol (IV) used for maintenance of general anesthesia
  Interventions: Diagnostic Test: Mini Mental State Examination(MMSE),Montreal Cognitive Assessment ( MoCA),S100B ( protein S100 subunit beta) ,GFAP ( glial fibrillary acidic protein ),NSE ( neuron-specific enolase )

INTERVENTIONS:
Diagnostic Test: Mini Mental State Examination(MMSE),Montreal Cognitive Assessment ( MoCA),S100B ( protein S100 subunit beta) ,GFAP ( glial fibrillary acidic protein ),NSE ( neuron-specific enolase ) — MMSE and MoCA will be applied preoperative,postoperative first day and fourth day S100B,GFAP and NSE will be measured in blood tests preoperative,postoperative second hour,postoperative 24. hour and postoperative 96. hour

SUMMARY:
Robotic assisted laparoscopic surgery has become an alternative to open or laparoscopic technique in various surgical fields. Robot assisted laparoscopic surgery is preferred by surgeons and patients due to easy accessibility, lower blood loss and lower transfusion rates. However, robotic assisted laparoscopic surgery can cause significant changes in cardiovascular, respiratory, metabolic and cerebral physiology because it requires a deep trendy position. When long -lasting deep trendelenburg position is applied, the cerebral autoregulation is impaired. In the literature, the presence of cases with brain edema is shown.

In recent years, many biomarkers have been used in the evaluation of brain damage. S100 Calcium Binding Protein (S100β), N Ron specific enolase (NSE), Glial Fibrils are among the biomarkers used to show acidic protein (GFAP) brain damage. The S100β is specific and is mainly produced by astrocytes and enters the bloodstream after neuron damage. Glial fibrils is an acidic protein (GFAP), a protein encoded by the GFAP gene in humans, an intermediate filament protein produced in the central nervous system. Neuron specific enolase (NSE) is one of the enzymes that increase brain damage encoded by Enolase 2 (ENO2) gene.

Mini Mental State Examination and Montreal Cognitive Assessment will be performed to determine neurological changes developing in patients.

The purpose of this study; Robotic assisted laparoscopic surgery is to examine the brain damage that may develop in patients due to deep trendelenburg position in patients with the said biomarkers and to evaluate the anesthesia methods applied in these surgery in line with the study results.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 18-75 who were operated on under general anesthesia for RALRP surgery and agreed to participate in the study will be included.

Exclusion Criteria:

* Participants who did not accept the study, had active intracranial pathology and history of intracranial pathology will not be included in the study.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients aged 18-75 who were operated on under general anesthesia for RALRP surgery
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-03-08 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
brain damage | in 96 hours
  Brain damge between the two groups will be compared

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz University Hospital, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Schramm P, Treiber AH, Berres M, Pestel G, Engelhard K, Werner C, Closhen D. Time course of cerebrovascular autoregulation during extreme Trendelenburg position for robotic-assisted prostatic surgery. Anaesthesia. 2014 Jan;69(1):58-63. doi: 10.1111/anae.12477. Epub 2013 Nov 20. PMID 24256501
- [Background] Amoo M, Henry J, O'Halloran PJ, Brennan P, Husien MB, Campbell M, Caird J, Javadpour M, Curley GF. S100B, GFAP, UCH-L1 and NSE as predictors of abnormalities on CT imaging following mild traumatic brain injury: a systematic review and meta-analysis of diagnostic test accuracy. Neurosurg Rev. 2022 Apr;45(2):1171-1193. doi: 10.1007/s10143-021-01678-z. Epub 2021 Oct 28. PMID 34709508